CLINICAL TRIAL: NCT04981301
Title: The Efficacy of Ultrasound-Guided Quadratus Lumborum Block for Pain Management Following Lumbar Spinal Surgery
Brief Title: Quadratus Lumborum Block for Lumbar Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 19
Record Dates: First submitted 2021-07-17; First posted 2021-07-28 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar Disc Herniation; Postoperative pain management; Quadratus Lumborum Block
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Ninety patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for lumbar disc herniation surgery will be included in the study. Patients will be randomly divided into two groups (Group Q = QLB group, Group C = Control group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Q = QLB group (Active Comparator): Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure.
  Interventions: Drug: Quadratus Lumborum Block
- Group C = Control group (No Intervention): Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure.
  Wound local anesthetic infiltration will be applied to the patients in the control group.

INTERVENTIONS:
Drug: Quadratus Lumborum Block — The block procedure will be applied after the surgery and before extubation with patients in the prone position by using US (Vivid Q, GE Healthcare, US). Under aseptic conditions using 10% povidone iodine, the convex probe will be covered with a sterile sheath and a 22G, 100 mm block needle (Braun Stimuplex Ultra 360, Germany) will be used. After visualizing the abdominal muscles with the anterior approach, the needle will be punctured in the Petit triangle and 5 ml of saline will be injected into the anterolateral border of the quadratus lumborum muscle. After the block location is confirmed, 15 ml of 0.25% bupivacaine will be injected. The same process will be applied to the opposite side (30 ml totally).
  Arms: Group Q = QLB group

SUMMARY:
Spine surgery in thoracolumbar region is one of the most common surgeries performed for the treatment of leg and back pain. Pain management is especially important for these patients since chronic pain often occurs after surgery. Severe pain may occur at postoperative period in patients following lumbar disc herniation (LDH) operation. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced.

Ultrasound-guided quadratus lumborum block (QLB) is a fascial plane block where local anesthetic is injected adjacent to the quadratus lumborum muscle with the goal of anesthetizing the thoracolumbar nerves.

The aim of this study is to evaluate the efficacy of US-guided QLB for postoperative analgesia management after lumbar disc herniation-laminectomy surgery. The primary aim is to evaluate postoperative pain scores (VAS), the secondary aim is to evaluate use of rescue analgesia and adverse effects (allergic reaction, nausea, vomiting).

DETAILED DESCRIPTION:
Spine surgery in thoracolumbar region is one of the most common surgeries performed for the treatment of leg and back pain. Pain management is especially important for these patients since chronic pain often occurs after surgery. Severe pain may occur at postoperative period in patients following lumbar disc herniation (LDH) operation. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced.

Opioids are one of the most preferred drugs among the analgesic agents. Parenteral opioids are generally performed for patients after surgery. However opioids have undesirable adverse events such as nausea, vomiting, itching, sedation and respiratory depression (opioid-related adverse events).

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment. US-guided interfascial plane blocks have been used increasily due to the advantages of ultrasound in anesthesia practice. Ultrasound-guided quadratus lumborum block (QLB) is a fascial plane block where local anesthetic is injected adjacent to the quadratus lumborum muscle with the goal of anesthetizing the thoracolumbar nerves.

The aim of this study is to evaluate the efficacy of US-guided QLB for postoperative analgesia management after lumbar disc herniation-laminectomy surgery. The primary aim is to evaluate postoperative pain scores (VAS), the secondary aim is to evaluate use of rescue analgesia and adverse effects (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for lumbar disc herniation surgery under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* Receiving anticoagulant treatment
* Known local anesthetics and opioid allergy
* Infection of the skin at the site of the needle puncture
* Pregnancy or lactation
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | Postoperative 24 hours period
  Change from Baseline Pain Scores at Postoperative 24 hours.

SECONDARY OUTCOMES:
The use of rescue analgesia | Postoperative 24 hours period
  Tramodol using

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Ueshima H, Otake H. RETRACTED: Clinical experience of anterior quadratus lumborum block after lumber surgery. J Clin Anesth. 2017 Feb;37:131. doi: 10.1016/j.jclinane.2016.12.014. Epub 2017 Jan 9. No abstract available. PMID 28235503 (Retraction: PMID 35393201 J Clin Anesth. 2022 Aug;79:110740)